CLINICAL TRIAL: NCT00908479
Title: Exercise Programs for Stroke: Effect of an Inpatient Supplementary Practice Program on Lower Extremity Function
Brief Title: The Effect of an Inpatient Home-work Exercise Program on Leg Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H09-00665
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Cerebrovascular Accident (Stroke)
Keywords: Exercise; Rehabilitation; leg function; in patient; RCT
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LE (Experimental): Leg Exercise group
  Interventions: Behavioral: Leg Exercise Program
- LM (Experimental): Leg Management (Control group)
  Interventions: Behavioral: Leg Management group

INTERVENTIONS:
Behavioral: Leg Exercise Program — Participants will engage in an extra 45-60 minutes per day of self-managed lower extremity homework exercises focused on improving strength, balance and walking ability.
  Other Names: Inpatient supplementary practice program on lower extremity function
  Arms: LE
Behavioral: Leg Management group — Therapist provides educational information about leg pain, recovery, bone density, and fall risk.
  Arms: LM

SUMMARY:
This study would focus on a new method of adding extra leg homework exercises to the usual therapy delivered in the hospital. We propose to design an exercise program for the affected leg that would be given to the client as homework and done in the client's hospital room or ward. The program would be designed and monitored by a therapist that works in the hospital.

DETAILED DESCRIPTION:
In total 120 participants admitted for stroke rehabilitation in the province British Columbia, Canada will be randomly assigned to either the Leg Exercise group or Leg Management group. The extra leg exercise group (experimental group) will receive usual therapy plus 60 minutes per day of self-directed leg exercises. This program will last for 4 weeks while the participant is in the hospital. The Leg Exercise program will include exercises of range of motion, leg strengthening, weight-bearing, and walking. The family will be encouraged to participate in the program with the participant. The control group (Leg Management group) will receive usual therapy and stroke education.

ELIGIBILITY:
Inclusion Criteria:

* Have been admitted to a hospital unit for stroke treatment
* 19 years or older
* Are experiencing difficulty using legs
* Able to understand and follow instructions

Exclusion Criteria:

* Have uncontrolled hypertension or unstable cardio-vascular condition
* Injuries to muscles, bones, or joints of the leg
* Unable to verbally speak or understand the investigators when asked questions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is gait speed | 4 weeks post-intervention

SECONDARY OUTCOMES:
The secondary outcomes will assess the effect of the experimental intervention on balance and physical activity | 4 weeks post-baseline, then 6 and 12 months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, Principal Investigator — University of British Columbia; William Miller, Study Director — University of British Columbia; Andrew Dawson, Study Director — University of British Columbia; Penny Brasher, Study Director — University of British Columbia
Locations (5):
- Canada (5):
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia
  - GF Strong Rehab Center, Vancouver, British Columbia
  - Holy Family Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia